CLINICAL TRIAL: NCT06277375
Title: Fibromiyalji Tanılı Kadınlarda Uygulanan Yavaş Vurumlu Sırt Masajının Ağrı ve Yorgunluk Üzerine Etkisi: Randomize Kontrolü Çalışma
Brief Title: The Effect of Slow Stroke Back Massage on Pain and Fatigue in Women With Fibromyalgia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Dilek Efe Arslan, ErciyesU, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 813/793
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Massage Intervention
Keywords: pain; Fatigue; Fibromyalgia
MeSH Terms: conditions — Pain; Fatigue; Fibromyalgia | interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow stroke back massage (Experimental): The application to the experimental group will be done 3 days a week for 10 minutes for a total of 30 minutes.
  Interventions: Behavioral: Massage
- Control Group (No Intervention): No intervation. Routine care.

INTERVENTIONS:
Behavioral: Massage — The application starts from the neck with small circular strokes with the thumbs. Surface strokes are performed with the palm of the hand from the base of the skull towards the sacral region. Then rhythmic strokes are repeated from the sacrum along the entire spine towards the skull.The application to the experimental group will be done 3 days a week for 10 minutes for a total of 30 minutes.
  Arms: Slow stroke back massage

SUMMARY:
Fibromyalgia syndrome (FM) is defined as a non-inflammatory chronic pain syndrome with widespread pain in the musculoskeletal system, tender points (PINs) on physical examination and no specific laboratory findings. T Sampling was calculated using Power power (G Power 3.1.9.4) analysis. The effect size of the study was calculated based on the mean pain scores and standard deviations of the control and experimental groups taken from the study conducted by Field, et al. (2002). Accordingly, when 25 patients were included in each group, it was determined that the power was 85% at 5% Type I error level. The application to the experimental group will be done 3 days a week for 10 minutes for a total of 30 minutes. data will be collected with patient information form, fatigue severity scale and vas.

DETAILED DESCRIPTION:
he research will be conducted experimentally with the aim of evaluating the effects of slow-stroke back massage in patients followed up in the physical therapy and rehabilitation unit with the diagnosis of fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate verbally,
* Over 18 years of age,
* no vision and hearing loss
* who have received medical treatment,
* who have never received a slow-stroke back massage before

Exclusion Criteria:

* Initially volunteered to participate in the study, but did not like the application of slow-stroke back massage
* who wants to leave the study for another reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
VAS | The scale was filled in the baseline
  VAS consisting of a 10-centimeter horizontal line, anchored evenly by numbers from 0 to 10, was used to assess the patient's pain and willingness to repeat the procedure. The number 0 was identical to having no pain while the number 10 corresponded to maximal pain that can be experienced by the patient.
Fatigue | The scale was filled in the baseline
  It is a tenitem, self-administered questionnaire. Because each item has a maximum possible score of 10, the maximum possible total score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK EFE ARSLAN, Study Director — ERCİYES UNİVERSİTY
Locations (1):
- Dilek Efe Arslan, Kayseri, Melikgazi, Turkey (Türkiye)